CLINICAL TRIAL: NCT01267305
Title: The Impact of Different Anticoagulant Therapy on Hemorrhage and Coagulation After Thoracic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Ming Zhong, department of anesthesiology and surgical intensive care unit, Shanghai Zhongshan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SICUTEG-01
Record Dates: First submitted 2010-12-25; First posted 2010-12-28 (Estimated); Last update posted 2014-04-29 (Estimated); Status verified 2014-04

CONDITIONS: Lung Neoplasms; Esophageal Neoplasms; Venous Thromboembolism
Keywords: esophagectomy; lung resection; venous thromboembolism; low molecular weight heparin; chest drainage; TEG
MeSH Terms: conditions — Lung Neoplasms; Esophageal Neoplasms; Venous Thromboembolism | interventions — Fondaparinux; Nadroparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- lung lmwh1 (Active Comparator): use LMWH once daily after lung resection
  Interventions: Drug: Nadroparin Calcium
- lung lmwh2 (Experimental): use LMWH twice daily after lung resection
  Interventions: Drug: Nadroparin Calcium
- lung Fondaparinux (Experimental): use Fondaparinux once daily after lung resection
  Interventions: Drug: Fondaparinux
- eso lmwh1 (Active Comparator): use LMWH once daily after esophagectomy
  Interventions: Drug: Nadroparin Calcium
- eso lmwh2 (Experimental): use LMWH twice daily after esophagectomy
  Interventions: Drug: Nadroparin Calcium
- eso Fondaparinux (Experimental): use Fondaparinux once daily after esophagectomy
  Interventions: Drug: Fondaparinux

INTERVENTIONS:
Drug: Fondaparinux — 2.5mg IH qd(8AM) after operation
  Other Names: ARIXTRA; H20080111
  Arms: eso Fondaparinux; lung Fondaparinux
Drug: Nadroparin Calcium — 4100AxaIU IH qd(8AM) after operation
  Other Names: Fraxiparine
  Arms: eso lmwh1; lung lmwh1
Drug: Nadroparin Calcium — 4100AxaIU IH q12h(8Am,8Pm) after operation
  Other Names: Fraxiparine
  Arms: eso lmwh2; lung lmwh2

SUMMARY:
The purpose of this study is to determine whether the use of different dose of LMWH compared with fondaparinux for thromboprophylaxis is efficacious and safety after thoracic surgery.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of esophageal carcinoma and planned for esophagectomy
* clinical diagnosis of lung carcinoma and planned for lung resection
* general anesthesia combined with epidural anesthesia

Exclusion Criteria:

* blood clotting disfunction before surgery
* anticoagulating or antiplatelet history before surgery
* low blood platelets count
* hemorrhagic disease
* cerebral hemorrhage
* cerebral,spinal,ophthalmologic operation history
* peptic ulcer
* bleeding>400ml in operation
* bleeding>100ml/h after operation
* blood transfusion in or after operation
* severe renal or liver disfunction
* severe hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 362 (Actual)
Dates: Start 2011-01; Primary Completion 2013-04 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
TEG values | three days after surgery
  1.5ml aterial blood sample will be obtained daily for TEG , and the vulues of TEG,such as R,K,Alpha angle,MA,G,CI ,will be measured

SECONDARY OUTCOMES:
bleeding quantity of chest drainage | three days after surgery
  all drain from chest tube are gathered and hematocrits are measured to calculate the quantities of bleeding
incidence rate of deep venous thromboembolism（DVT) | after surgery up to 7 days
  incidence of DVT is measured by vascular ultrasonography
inhospital mortality | after surgery up to 28 days
  the number of death in the period of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Lizhen Xuan, Principal Investigator — Shanghai Zhongshan Hospital
Locations (1):
- Zhongshan Hospital, Shanghai, China